CLINICAL TRIAL: NCT06552143
Title: An Applied Study on the Use of Stone Needles Therapy to Assist the Rehabilitation of Maternal Diastasis Rectus Abdominis Based on the Theory of Belt Channel
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yunnan University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Zuoqin Zhang, Graduate Nursing Students, Yunnan University of Chinese Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XW2023-025
Record Dates: First submitted 2024-07-24; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Diastasis Recti Abdominis
Keywords: postpartum diastasis rectus abdominis Belt channel; stone needle therapy; Belt channel; rehabilitative nursing

STUDY DESIGN:
Intervention Model Description: The patients were divided into control and intervention groups according to the time of their visit to the clinic. The patients who met the inclusion and exclusion criteria of the study from February to May 2023 were the control group and the patients who met the inclusion and exclusion criteria of the study from June to September 2023 were the intervention group. The number of patients in each group was 60.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor did not know whether the patient being measured belonged to the control or intervention group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stone needle therapy follows the Belt channel (Other): generic name: Stone needle therapy frequency: Neuromuscular Electrical Stimulation (NMES) for a total of 10 sessions, with the addition of massage therapy after the 3rd, 6th, and 9th NMES sessions, and stone needle therapy after each massage session for a total of 3 sessions.
  dosage: Thirty minutes at a time, three times in total.
  Interventions: Other: Stone needle therapy follows the Belt channel
- control group (Other): generic name: Neuromuscular Electrical Stimulation combined with massage therapy frequency: Neuromuscular Electrical Stimulation (NMES) for a total of 10 sessions, with the addition of massage therapy after the 3rd, 6th, and 9th NMES sessions.
  dosage: Thirty minutes at a time, three times in total.
  Interventions: Other: Stone needle therapy follows the Belt channel

INTERVENTIONS:
Other: Stone needle therapy follows the Belt channel — Stone needle therapy follows the Belt channel involves the use of stones by the intervener to follow the path of the Belt channel by pushing and rubbing the abdomen of patients with postpartum diastasis rectus abdominis.

SUMMARY:
This clinical trial aims to find out whether stone needles therapy can effectively assist in the treatment of maternal diastasis rectus abdominis (DRA) based on the Belt channel theory, it will also validate whether the Ben-Tovim Walker body attitude questionnaire (BAQ) can be used as a tool to measure body image satisfaction in Chinese patients with postpartum DRA. The main questions it aims to answer are: Can stone needles therapy promote the recovery of maternal DRA? Whether the Chinese version of the Body attitude questionnaire (BAQ-C) can be used as a body image satisfaction measurement tool for patients with postpartum DRA. The researchers will add stone needles therapy to neuromuscular electrical stimulation (NMES) and massage therapy to see if stone needles therapy can promote the recovery of postpartum DRA.

DETAILED DESCRIPTION:
Participants will: Receive NMES combined with massage therapy or the addition of stone needles therapy on a sub-basis every day for 10 days.

Abdominal circumference, inner rectus distance will be measured and recorded after each treatment Body imagery satisfaction, low back pain and dysfunction scores, anxiety, depression scores, and quality of life scores will be measured after all treatments are completed.

ELIGIBILITY:
Inclusion Criteria:

1. patients who meet the diagnostic criteria of postpartum rectus abdominis muscle separation, and the distance of rectus abdominis muscle separation is ≥3.0cm with postpartum low back pain.
2. Patients who are >42d postpartum and have cleaned up their discharge;
3. Women who are 42day-3 mouths after normal delivery;
4. Postpartum women who have not received any other treatment before treatment in our hospital;

Exclusion Criteria:

1. With severe parenchymal organ diseases such as renal, cardiac, or hepatic diseases or due to comorbid cognitive impairment, Alzheimer's disease or psychological or psychiatric diseases can not complete the cooperation, etc;
2. Those with contraindications to stone therapy;
3. Those with contraindications to bioelectric stimulation therapy.
4. Combined with puerperal infection and gastrointestinal adhesion;
5. Patients with postpartum back pain due to other reasons such as lumbar disc herniation or kidney stones;
6. Patients who cannot tolerate the program;

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
inter-recti distance | pre-intervention and after three stone needle therapies interventions
  Bilateral rectus abdominis distance
Abdominal circumference | pre-intervention and after three stone needle therapies interventions
  Horizontal circumference of the abdomen via the iliac crest point.
Body Image Satisfaction | pre-intervention and after intervention
  Body image satisfaction refers to how a person perceives, thinks, or feels about his or her body.

SECONDARY OUTCOMES:
Low back pain Visual Analogue Scale | pre-intervention and after intervention
  A 10 cm horizontal line is drawn on top of the paper, and the visual analogue scale (VAS) is used for the horizontal line. The line is 0mm at one end, which means 'no pain at all'; 10mm at the other end, which means 'extreme pain'; the pain level increases from 0mm to 10mm, with higher scores representing more intense pain.
Oswestry Disability Index | pre-intervention and measured immediately after completion of all treatments
  The Oswestry Disability Index (ODI) is a widely used measure for assessing the function a limitations and disability associated with lower back pain. This index provides a standardized way to evaluate the impact of back pain on a person's daily activities and overall quality of life.
Self-Rating Anxiety Scale | pre-intervention and measured immediately after completion of all treatments
  It is a commonly used psychometric tool developed by the American psychologist Zung, and is a self-report scale used to assess an individual's level of anxiety.
Edinburgh postnatal depression scale | pre-intervention and measured immediately after completion of all treatments
  A standardized questionnaire to detect symptoms of depression in postnatal women.
THE WORLD HEALTH ORGANIZATION QUALITY OF LIFE | pre-intervention and measured immediately after completion of all treatments
  It is a tool used to assess people's quality of life, which helps to collect and analyse information about the individual's state of health, psychological functioning, social competence, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, Principal Investigator — The First Affiliated Hospital of Yunnan University of Chinese Medicine
Locations (1):
- YunNan Provincial Hospital of Traditional Chinese Medicine, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No